CLINICAL TRIAL: NCT02216578
Title: Phase II Study of Cabozantinib in Patients With Gastrointestinal Stromal Tumor (GIST) Who Progressed During Neoadjuvant, Adjuvant or Palliative Therapy With Imatinib and Sunitinib
Brief Title: Ph II CABOGIST in GIST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1317; 2014-000501-13 (EudraCT Number)
Record Dates: First submitted 2014-07-31; First posted 2014-08-15 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Gastrointestinal Stromal Tumor
Keywords: tyrosine kinase inhibitor; progressed; (GIST)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cabozantinib (Experimental): cabozantinib 60 mg oral daily
  Interventions: Drug: cabozantinib

INTERVENTIONS:
Drug: cabozantinib — Oral

SUMMARY:
The study is a multi-center, multi-national, open label, single arm Phase II study of single-agent cabozantinib. The objective of the study is to assess the safety and activity of cabozantinib in patients with metastatic GIST who have previously progressed on imatinib and sunitinib and have not been exposed yet to other KIT- or PDGFR-directed tyrosine kinase inhibitors.

Patient will receive cabozantinib until they experience no further benefit from the treatment, becoming intolerant to the drug or wishing to discontinue the treatment. Treatment beyond RECIST 1.1 progression is allowed in patients deriving clinical benefit upon investigator's discretion, provided no other criteria for treatment withdrawal are met.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of GIST that is metastatic. Patients with the primary tumor still in place are excluded from the trial, due to the risk for intestinal perforation reported for cabozantinib.
* Presence of at least one non-previously irradiated, measurable metastatic lesion as defined by RECIST 1.1.
* Archival tumor tissue available from primary tumor or metastatic site (10 unstained slides with archived tumor tissue of 10 micrometer thickness and two hematoxylin and eosin (H&E) stained slides) for central mutational analysis; Note: slides are preferred material but if not available blocks are accepted
* Failure on prior therapy with

  * Interval from prior TKI therapy to the first dose of cabozantinib should be at least 14 days
  * Radiological progression on imatinib during neoadjuvant, adjuvant or palliative treatment of GIST or within 3 months after completing adjuvant treatment with imatinib AND radiological progression on sunitinib for the treatment of advanced GIST

Note: progression is assessed by local radiologist/oncologist without central confirmation of pre-baseline progression.

* Agreement of the patient to allow sequential sampling of circulating cell-free DNA for central mutational analysis is mandatory.
* Male or female patient ≥ 18 years of age
* ECOG (Eastern Cooperative Oncology Group) performance status (PS) of 0-1
* Adequate bone marrow and organ function as defined by the following laboratory values assessed within ≤ 14 days prior to receiving the first dose of study treatment:

  * ANC (Absolute Count Neutrophils) ≥ 1.5 x 10exp9/L (no prophylactic administration of G-CSF (Granulocyte Colony Stimulating Factor) or GM (Granulocyte Macrophage) -CSF allowed).
  * Platelet count ≥ 100 x 10exp9/L or x 10exp3/μL (transfusion allowed).
  * Hemoglobin ≥ 9.0 g/dL or 5.6 mmol/L (transfusion and erythropoietin allowed).
  * Prothrombin time (PT)/ INR (International Normalized Ratio) or partial thromboplastin time (PTT) test < 1.3 X ULN within 7 days before the first dose of study treatment; Note: patients requiring concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (eg, clopidogrel) are not eligible. Low dose aspirin (≤ 81 mg/day), low-dose warfarin (≤ 1 mg/day), and prophylactic LMWH (Low Molecular Weight Heparin) are permitted;
  * Potassium, calcium, magnesium and phosphorous within normal limits of the institution or corrected to within normal limits prior to the first dose of study medication.
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min or GFR >30 mL/min (as assessed per local standard).
  * Serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with Gilbert's syndrome).
  * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within ≤ 3.0 x ULN.
  * Serum albumin ≥ 2.8 g/dL.
  * Serum lipase < 2 x ULN and no radiologic or clinical evidence of pancreatitis
  * Urine protein/creatinine ratio (UPCR) ≤ 1.
* Clinically normal cardiac function based on the institutional lower limit of normal for left ventricular ejection fraction as assessed either by multi-gated acquisition scan or cardiac ultrasound, 12 lead ECG without clinically relevant abnormalities (stable atrial fibrillation allowed), no history of congenital long QT syndrome, no prolongation of corrected QT interval (QTcF) > 500 msec according to Fridericia's formula), and no history of any one of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting.
  * Myocardial infarction.
  * Unstable angina.
  * Coronary artery bypass graft surgery.
  * Clinically significant cardiac arrhythmias
  * Symptomatic peripheral vascular disease.
  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA).
* Patients must be able to swallow and retain oral film-coated tablets.
* Recovery to baseline or ≤ Grade 1 CTCAE v.4.0 from toxicities related to any prior treatments, unless AE(s) are clinically non significant and/or stable on supportive therapy;
* Prior surgery:

  * Minor surgery (including uncomplicated tooth extractions) within 28 days before the first dose of study treatment with complete wound healing at least 10 days before the first dose of study treatment is permitted.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the first dose of study treatment.

Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (ie, females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.

* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 4 months after the last study treatment. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Before patient registration, written informed consent must be given according to ICH (International Conference on Harmonisation)/GCP (Good clinical Practice), and national/local regulations.

Exclusion Criteria:

* evidence of tumor invading the gastrointestinal tract (esophagus, stomach, small or large bowel, rectum or anus) within 28 days prior to the first dose of cabozantinib.
* current evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib.
* radiographic presence of a cavitating pulmonary lesion within 28 days prior to the first dose of cabozantinib. patient with tumor in contact with, invading or encasing a major blood vessel
* other prior tyrosine kinase inhibitors for the treatment of advanced GIST.
* other investigational agents within 28 days before the first dose of study treatment;
* specific contraindications for treatment with cabozantinib (e.g. no known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to cabozantinib).
* poorly controlled hypertension defined at baseline as blood pressure (BP) >150/90 mmHg.
* cerebrovascular accident, no transient ischemic attack and no pulmonary embolism in the past 6 months.
* gastrointestinal disorders associated with a high risk of perforation or fistula formation within 28 days before the first dose of study treatment, including the following:

  * Known intra-abdominal tumor/metastases invading gastrointestinal mucosa.
  * Active peptic ulcer disease.
  * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis.
  * Malabsorption syndrome.
* One of the following within 6 months before the first dose of study treatment:

  * Clinically significant gastrointestinal bleeding.
  * Abdominal fistula.
  * Gastrointestinal perforation.
  * Bowel obstruction.
  * Gastric outlet obstruction.
  * Intra-abdominal abscess (complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment).
* other disorders associated with a high risk of fistula formation including PEG tube placement within 3 months before the first dose of study therapy;
* evidence of significant active bleeding (including GI bleeding) or bleeding diathesis within 6 months before the first dose of study treatment.
* hemoptysis ≥ 0.5 teaspoon (2.5 ml) of red blood within 3 months before the first dose of study treatment.
* signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment.

Note: patient with a prior history of hemoptysis associated with metastatic disease must have a bronchoscopy to rule out endobronchial lesions. A patient with an endobronchial tumor lesion is not eligible for the study.

* Prior surgery:

  * prior major surgery or trauma within 12 weeks prior to first dose of study drug and/or presence of any non-healing wound, fracture or ulcer. Complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment.
  * Patients with clinically relevant ongoing complications from prior surgery;
* Following clinically significant disorders such as:

  * active infection requiring systemic treatment within 28 days before the first dose of study treatment;
  * history of organ transplant;
  * concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment.
* history of other malignancy in the past 5 years with the exception of treated carcinoma in situ of the cervix and non-metastatic, non-melanoma skin cancer. Patients with desmoid fibromatosis or neurofibromas, which can be associated with GIST, are allowed to enter the trial, under the provision that they do have a measurable GIST lesion that can be distinguished from the other lesions.
* Patients requiring chronic concomitant treatment with strong CYP3A4 inducers (eg, dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's Wort)
* Lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | at 12 weeks

SECONDARY OUTCOMES:
Progression Free Survival (PFS) (RECIST 1.1) | at 12 weeks
  assessed with independent central review of radiological images
Overall survival (OS) | at 12 weeks
Objective response rate (ORR), defined as Complete Response (CR)+ Partial Response (PR) (RECIST 1.1) | 3 years
  assessed with independent central review of radiological images
Clinical benefit rate (CBR) defined as CR+PR+ SD (Stable Disease) (RECIST 1.1) | 3 years
  assessed with independent central review of radiological images.
Time to treatment failure (TTF) | 3 years
  Time to treatment failure (TTF) defined as treatment beyond progression is allowed by the protocol at the discretion of the treating physician)
Occurence of adverse events | 3 years
  Safety will be graded according to the Common Terminology Criteria (CTC) for Adverse Events (AE), CTC-AE version 4.0

OTHER OUTCOMES:
mutational subtypes of GIST | 3 years
  Prevalence of different mutational subtypes of GIST in archived tumor material derived from the primary tumor or a metastatic site and relative efficacy of cabozantinib in recruited mutational subsets
circulating plasma DNA | 3 years
  Feasibility of using circulating plasma DNA as "liquid biopsy" for mutational analysis in metastatic GIST with assessment of the concordance of results with conventional tissue-based mutational analysis

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schöffski, MD, Principal Investigator — U.Z. Leuven -Campus Gasthuisberg, Leuven, Belgium
Locations (11):
- U.Z. Leuven - Campus Gasthuisberg (147), Leuven, Belgium
- University Hospital Motol (1905), Prague, Czechia
- France (3):
  - Institut Bergonie (228), Bordeaux
  - Centre Leon Berard (227), Lyon
  - Gustave Roussy (225), Villejuif
- UniversitaetsMedizin Mannheim (527), Mannheim, Germany
- Military Hospital - State Health Centre (3769), Budapest, Hungary
- United Kingdom (4):
  - Clatterbridge Centre for Oncology NHS Trust - Clatterbridge Cancer Centre NHS Foundation Trust (659), Bebington
  - Royal Marsden Hospital - Chelsea, London (613), Chelsea
  - University College London Hospitals NHS Foundation Trust - University College Hospital (622), London
  - The Christie NHS Foundation Trust (610), Manchester

REFERENCES:
- [Derived] Kyriazoglou A, Jespers P, Vandecavaye V, Mir O, Kasper B, Papai Z, Blay JY, Italiano A, Zaffaroni F, Litiere S, Nzokirantevye A, Schoffski P. Exploratory analysis of tumor imaging in a Phase 2 trial with cabozantinib in gastrointestinal stromal tumor: lessons learned from study EORTC STBSG 1317 'CaboGIST'. Acta Oncol. 2022 Jun;61(6):663-668. doi: 10.1080/0284186X.2022.2068967. Epub 2022 Apr 28. PMID 35481400
- [Derived] Schoffski P, Mir O, Kasper B, Papai Z, Blay JY, Italiano A, Benson C, Kopeckova K, Ali N, Dileo P, LeCesne A, Menge F, Cousin S, Wardelmann E, Wozniak A, Marreaud S, Litiere S, Zaffaroni F, Nzokirantevye A, Vanden Bempt I, Gelderblom H. Activity and safety of the multi-target tyrosine kinase inhibitor cabozantinib in patients with metastatic gastrointestinal stromal tumour after treatment with imatinib and sunitinib: European Organisation for Research and Treatment of Cancer phase II trial 1317 'CaboGIST'. Eur J Cancer. 2020 Jul;134:62-74. doi: 10.1016/j.ejca.2020.04.021. Epub 2020 May 26. PMID 32470848